CLINICAL TRIAL: NCT05023161
Title: Non-invasive Prenatal Testing of Placental Chromosomal Abnormalities in Fetus With Intrauterine Growth Restriction
Brief Title: Non-invasive Placental Chromosome Exploration of Intrauterine Growth Restriction
Acronym: DPNI-RCIU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/12
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Fetal Growth Retardation
Keywords: Non Invasive Prenatal Testing; cell- free DNA; trisomy; placenta confined mosaic
MeSH Terms: conditions — Fetal Growth Retardation; Trisomy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient having a fetus with intra-uterine growth restriction diagnosis below the 3rd percentile
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Performed a 10 ml blood sample in each of the 200 patients included.

SUMMARY:
The objective of this project is the non-invasive prenatal detection of placenta-limited aneuploidies, in patients whose fetuses have a intrauterine growth restriction below 3rd percentile, in parallel with an amniocentesis.

This study will allow the chromosomal study of the placenta in pregnant women whose genetic prenatal diagnosis, made by amniocentesis, does not allow exploring the placental causes of fetal RCIU.

DETAILED DESCRIPTION:
Placental chromosomal aneuploidies will be detected by high-throughput whole genome sequencing of non-cellular DNA present in maternal plasma during pregnancy.

The study of the cfDNA will be carried out from a blood sample with the automated solution VERISEQ NIPT (Illumina) using the software illumina VeriSeq v2, allowing the detection of all chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* treated in the DDIANE fetal medicine centre at the Bordeaux University Hospital,
* having a fetus with IUGR diagnosis below the 3rd percentile (after reference medical ultrasound),
* from 16 weeks of amenorrhea or more,
* accepting an Invasive Prenatal Diagnosis by amniocentesis with array comparative genomic hybridization

Exclusion Criteria:

Childbearing women who:

* do not accept a non-invasive prenatal diagnosis (amniocentesis)
* have a fetus with non-isolated IUGR (associated with other ultrasound signs)
* do not consent to participate in the research protocol

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — having a fetus with IUGR diagnosis below the 3rd percentile (after reference medical ultrasound)
Study Population: Patient having a fetus with IUGR diagnosis below the 3rd percentile (after reference medical ultrasound)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-10-05 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Determine the presence or absence of chromosomal abnormality in the plasma sample. studied. | Inclusion date
  The result will be expressed in presence or absence of chromosomal abnormality such as trisomy, monosomy, deletion or duplication. The result will be compared with the fetal chromosome analysis carried out concomitantly on liquid amniotic as part of the treatment: if the analysis on Liquid Amniotic shows the same anomaly, it means that it is a fetal abnormality, if the Liquid Amniotic test is normal, it means that it is most likely an abnormality placental chromosome.

SECONDARY OUTCOMES:
Determine the proportion of chromosomal placental etiology in Intrauterine Growth Restriction. | Inclusion date
  Proportion will be described in terms of percentage counts and 95% confidence interval depending on the test Fisher's exact (p <0.05)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hôpital Antoine Béclère, Clamart
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No